CLINICAL TRIAL: NCT00115765
Title: PACCE: A Randomized, Open-Label, Controlled, Clinical Trial of Chemotherapy and Bevacizumab With and Without Panitumumab in the First-Line Treatment of Subjects With Metastatic Colorectal Cancer
Brief Title: PACCE: Panitumumab Advanced Colorectal Cancer Evaluation Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20040249
Record Dates: First submitted 2005-06-26; First posted 2005-06-27 (Estimated); Results first posted 2010-09-14 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-09

CONDITIONS: Colorectal Cancer
Keywords: Panitumumab Advanced Colorectal Cancer Evaluation Study (PACCE Study); Colorectal, Colon, Rectal Cancer, Metastatic Colorectal; Cancer; EGFr, Clinical Trial; Panitumumab, ABX-EGF; Immunex, Abgenix, Amgen; Metastatic Colorectal Cancer; Oncology
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms; Neoplasms | interventions — Oxaliplatin; Panitumumab; IFL protocol; Bevacizumab

ARMS (4):
- Oxaliplatin and bevacizumab without panitumumab (Active Comparator): Oxaliplatin-based chemotherapy and Bevacizumab Q2W alone.
  Interventions: Drug: Oxaliplatin Based Chemotherapy; Drug: Bevacizumab
- Irinotecan and bevacizumab plus panitumumab (Experimental): Irinotecan-based chemotherapy and Bevacizumab Q2W plus panitumumab 6mg/kg Q2W
  Interventions: Drug: Panitumumab; Drug: Irinotecan Based Chemotherapy; Drug: Bevacizumab
- Irinotecan and bevacizumab without panitumumab (Active Comparator): Irinotecan-based chemotherapy and Bevacizumab Q2W alone
  Interventions: Drug: Irinotecan Based Chemotherapy; Drug: Bevacizumab
- Oxaliplatin and bevacizumab plus panitumumab (Experimental): Oxaliplatin-based chemotherapy and Bevacizumab Q2W plus panitumumab 6mg/kg Q2W
  Interventions: Drug: Oxaliplatin Based Chemotherapy; Drug: Panitumumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: Oxaliplatin Based Chemotherapy — Oxaliplatin-based Chemotherapy Every 2 Week Regimens (Q2W Cycles) consisting of Oxaliplatin, Leucovorin (LV), 5-Fluorouracil (5-FU) - To be determined by physician. On Day 1 irinotecan and LV are given at the same time using different bags and a Y-line followed by 5-FU administration.
  Other Names: FOLFOX 4; FOLFOX 5; Modified FOLFOX 6; FOLFOX 7; Oxaliplatin
  Arms: Oxaliplatin and bevacizumab plus panitumumab; Oxaliplatin and bevacizumab without panitumumab
Drug: Panitumumab — PanitumumabPanitumumab is a high affinity (Kd = 5 x 10-11 M) fully human IgG2 monoclonal antibody that is directed against the human EGFr. Panitumumab will be administered by a 30-60 minute IV infusion at a dose of 6 mg/kg once every 2 weeks on the same day of the oxaliplatin- or irinotecan-based chemotherapy and bevacizumab.
  Other Names: pmab; Vectibix
  Arms: Irinotecan and bevacizumab plus panitumumab; Oxaliplatin and bevacizumab plus panitumumab
Drug: Irinotecan Based Chemotherapy — Irinotecan-based Chemotherapy Every 2 Week Regimens (Q2W Cycles) - Irinotecan, Leucovorin (LV), 5-Fluorouracil (5-FU) - To be determined by physician. On Day 1 irinotecan and LV are given at the same time using different bags and a Y-line followed by 5-FU administration.
  Other Names: FOLFIRI; Douillard
  Arms: Irinotecan and bevacizumab plus panitumumab; Irinotecan and bevacizumab without panitumumab
Drug: Bevacizumab — Bevacizumab is a vascular endothelial growth factor (VEGF)-targeted antibody therapy that was administered to subjects intravenously Q2 weeks as per usual standard of care on the same day of chemotherapy and panitumumab administration .
  Other Names: Avastin

SUMMARY:
The purpose of this study is to assess whether treatment with the study drug, panitumumab given concomitantly with every 2 (Q2) week oxaliplatin-based chemotherapy and bevacizumab improves progression-free survival (PFS) compared to treatment Q2-week with oxaliplatin-based chemotherapy and bevacizumab alone. All subjects will receive Q2-week oxaliplatin- or irinotecan-based chemotherapy and bevacizumab. Control arm subjects will not receive concomitant panitumumab therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the colon or rectum
* Metastatic colorectal cancer (mCRC)
* Measurable disease per modified response evaluation criteria in solid tumors (RECIST) criteria
* ECOG performance status of 0 or 1
* Available paraffin-embedded tumor tissue (from primary tumor or metastasis) or unstained slides of paraffin-embedded tissue
* If history of other primary cancer, subject will be eligible only if she or he has:

  * Curatively resected non-melanomatous skin cancer;
  * Curatively treated cervical carcinoma in situ;
  * Other primary solid tumor curatively treated with no known active disease present and no treatment administered for the last 5 years.
* Adequate hematologic data as follows:

  * Absolute neutrophil count (ANC) greater than or equal to 1.5 x 10^9 cells/L;
  * Platelet count greater than or equal to 100 x 10^9/L;
  * Hemoglobin greater than or equal to 9.0 g/dL. - Adequate renal function:
  * Serum creatinine less than or equal to 1.5 x upper limit of normal (ULN);
  * Urinary protein dipstick of less than 2+ (if urinary dipstick 2+ or greater, then excretion of less than or equal to 1000 mg of protein per day as determined by 24-hour urine collection).
* Adequate hepatic function:

  * Alkaline phosphatase less than or equal to 3 x ULN (if liver metastases, less than or equal to 5 x ULN);
  * Aspartate aminotransferase (serum glutamic-oxaloacetic transaminase)(AST) less than or equal to 3 x ULN (if liver metastases, less than or equal to 5 x ULN);
  * Alanine aminotransferase (serum glutamic-pyruvic transaminase) (ALT) less than or equal to 3 x ULN (if liver metastases, less than or equal to 5 x ULN);
  * Bilirubin less than or equal to 2 x ULN. - Competent to comprehend, sign, and date an IRB-approved informed consent form
* Before any study-specific procedure, the appropriate written informed consent must be obtained.

Exclusion Criteria:

* Prior chemotherapy or biologic (i.e., antibody or vaccine) treatment for mCRC disease - Last dose of adjuvant or radiosensitizing chemotherapy less than 6 months before randomization - Radiotherapy within 14 days before randomization
* Elective and/or planned major surgical procedure to be performed during the course of this trial (surgery that arises as needed or necessary during the course of the study, not agreed a priori, will not make the subject ineligible)
* Major surgery within 28 days before randomization
* Central nervous system metastases
* History of interstitial pneumonitis or pulmonary fibrosis or evidence of interstitial pneumonitis or pulmonary fibrosis on baseline chest X-ray or CT-scan
* Clinically significant ascites
* Preexisting bleeding diathesis or coagulopathy or the need for full-dose anticoagulation
* Any of the following within 1 year before randomization:

  * Myocardial infarction;
  * Unstable angina;
  * Symptomatic congestive heart failure;
  * Serious uncontrolled cardiac arrhythmia;
  * Cerebrovascular accident or transient ischemic attack;
  * Gastrointestinal ulcer or hemorrhage;
  * Hemoptysis;
  * Pulmonary embolism;
  * Deep vein thrombosis, or other significant thromboembolic event.
* Regular use of non-steroidal anti-inflammatory agents
* Female subject of childbearing potential, not abstinent, and not willing to use contraceptives during the course of the study and for 6 months following the last dose of first-line treatment
* Female subject who is breast-feeding or who has positive serum pregnancy test 72 hours prior to randomization
* Male subject, not abstinent, and not willing to use adequate contraception upon enrollment into this study and for 6 months following the last dose of first-line treatment
* Subject known to be human immunodeficiency virus (HIV) positive
* Subject allergic to panitumumab or any components of panitumumab formulation
* History of any medical or psychiatric condition or laboratory abnormality that, in the opinion of the investigator, may increase the risks associated with study participation or study drug administration or may interfere with the conduct of the study or interpretation of study results
* Subject unwilling or unable to comply with study requirements
* Any kind of disorder that compromises the ability of the subject to give written informed consent and/or comply with the study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1053 (Actual)
Dates: Start 2005-06-01 (Actual); Primary Completion 2007-05-31 (Actual); Study Completion 2009-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Hecht JR, Mitchell E, Chidiac T, Scroggin C, Hagenstad C, Spigel D, Marshall J, Cohn A, McCollum D, Stella P, Deeter R, Shahin S, Amado RG. A randomized phase IIIB trial of chemotherapy, bevacizumab, and panitumumab compared with chemotherapy and bevacizumab alone for metastatic colorectal cancer. J Clin Oncol. 2009 Feb 10;27(5):672-80. doi: 10.1200/JCO.2008.19.8135. Epub 2008 Dec 29. PMID 19114685
- [Derived] Abdel-Rahman O. Effect of Body Mass Index on 5-FU-Based Chemotherapy Toxicity and Efficacy Among Patients With Metastatic Colorectal Cancer; A Pooled Analysis of 5 Randomized Trials. Clin Colorectal Cancer. 2019 Dec;18(4):e385-e393. doi: 10.1016/j.clcc.2019.07.005. Epub 2019 Jul 15. PMID 31378656
- [Derived] Abdel-Rahman O. Impact of Sex on Chemotherapy Toxicity and Efficacy Among Patients With Metastatic Colorectal Cancer: Pooled Analysis of 5 Randomized Trials. Clin Colorectal Cancer. 2019 Jun;18(2):110-115.e2. doi: 10.1016/j.clcc.2018.12.006. Epub 2018 Dec 28. PMID 30679026
- See also: FDA-approved Drug Labeling — http://www.vectibix.com/
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 10 March 2005 through 19 October 2006.
Groups:
- Oxaliplatin and Bevacizumab Plus Panitumumab: Oxaliplatin-based chemotherapy and Bevacizumab Q2W plus panitumumab 6 mg/kg Q2W
- Irinotecan and Bevacizumab Plus Panitumumab: Irinotecan-based chemotherapy and Bevacizumab Q2W plus panitumumab 6 mg/kg Q2W
Period: Overall Study
Arm/Group | Irinotecan and Bevacizumab Without Panitumumab | Oxaliplatin and Bevacizumab Plus Panitumumab | Oxaliplatin and Bevacizumab Without Panitumumab | Irinotecan and Bevacizumab Plus Panitumumab
Started | 115 | 413 | 410 | 115
Completed | 80 (Participants who were on study at closure or died) | 313 (Participants who were on study at closure or died) | 289 (Participants who were on study at closure or died) | 84 (Participants who were on study at closure or died)
Not Completed | 35 | 100 | 121 | 31
Not completed — Withdrawal by Subject | 22 | 53 | 76 | 15
Not completed — Physician Decision | 4 | 15 | 18 | 13
Not completed — Lost to Follow-up | 3 | 20 | 18 | 1
Not completed — Other | 6 | 12 | 9 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxaliplatin and Bevacizumab Without Panitumumab | Irinotecan and Bevacizumab Plus Panitumumab | Irinotecan and Bevacizumab Without Panitumumab | Oxaliplatin and Bevacizumab Plus Panitumumab | Total
Number analyzed (Participants) | 410 | 115 | 115 | 413 | 1053
Age, Continuous [Mean (Standard Deviation); unit: Year] | 61.0 (11.9) | 59.4 (11.7) | 57.8 (12.0) | 60.8 (11.7) | 60.4 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 172 | 59 | 44 | 180 | 455
  Male | 238 | 56 | 71 | 233 | 598
Race/Ethnicity, Customized [Number; unit: Participant]
  White or Caucasian | 330 | 86 | 85 | 343 | 844
  Black or African American | 41 | 18 | 16 | 35 | 110
  Hispanic or Latino | 25 | 6 | 14 | 25 | 70
  Asian | 10 | 2 | 0 | 10 | 22
  Japanese | 2 | 0 | 0 | 0 | 2
  American Indian or Alaska Native | 1 | 2 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Other | 0 | 1 | 0 | 0 | 1
ECOG Score [Number; unit: Participant] — Eastern Cooperative Oncology Group (ECOG) Score
  Participant
    0 | 239 | 68 | 74 | 253 | 634
    1 | 171 | 47 | 41 | 160 | 419
Number of Metastatic Organs [Number; unit: Participant]
  None | 0 | 0 | 0 | 1 | 1
  1 | 199 | 46 | 53 | 204 | 502
  >1 | 211 | 69 | 62 | 208 | 550
Primary Site of Disease [Number; unit: Participant]
  Colon | 326 | 92 | 95 | 322 | 835
  Rectal | 84 | 23 | 20 | 91 | 218
Prior adjuvant chemotherapy [Number; unit: Participant]
  Yes | 77 | 38 | 36 | 80 | 231
  No | 333 | 77 | 79 | 333 | 822

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (Oxaliplatin)
Description: Kaplan-Meier estimate of the median time from randomization to death from any cause or first observed disease progression
Time Frame: Overall study
Population: Intention-to-Treat
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | Oxaliplatin and Bevacizumab Plus Panitumumab | Oxaliplatin and Bevacizumab Without Panitumumab
Number analyzed (Participants) | 413 | 410
Month | 10.0 [8.9 to 11.0] | 11.4 [10.5 to 11.9]
Statistical Analysis 1: Comparison: Oxaliplatin and Bevacizumab Plus Panitumumab vs Oxaliplatin and Bevacizumab Without Panitumumab; Test type: Superiority or Other; p = 0.011, Regression, Cox; Model covariates were ECOG status, prior chemotherapy, metastatic organs, disease site, oxaliplatin dose < 85 mg/m2, and oxaliplatin dose > 100 mg/m2; Hazard Ratio (HR) = 1.27, 95% CI [1.06 to 1.52]

2. Secondary Outcome: Overall Survival (Oxaliplatin)
Description: Kaplan-Meier estimate of the median time from randomization to death from any cause in groups treated with Oxaliplatin
Time Frame: Overall study
Population: Intention-to-Treat
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | Oxaliplatin and Bevacizumab Plus Panitumumab | Oxaliplatin and Bevacizumab Without Panitumumab
Number analyzed (Participants) | 413 | 410
Month | 19.4 [18.4 to 20.8] | 24.5 [20.4 to 24.5]
Statistical Analysis 1: Comparison: Oxaliplatin and Bevacizumab Plus Panitumumab vs Oxaliplatin and Bevacizumab Without Panitumumab; Test type: Superiority or Other; p = 0.005, Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.43, 95% CI [1.11 to 1.83]

3. Secondary Outcome: Objective Tumor Response Rate (Oxaliplatin)
Description: Best overall response of complete or partial response within oxaliplatin stratum
Time Frame: Overall study
Population: Intention-to-Treat
Measure: Number; unit: Participant
Arm/Group | Oxaliplatin and Bevacizumab Plus Panitumumab | Oxaliplatin and Bevacizumab Without Panitumumab
Number analyzed (Participants) | 413 | 410
Participant | 190 | 196

4. Secondary Outcome: Time to Progression (Oxaliplatin)
Description: Kaplan-Meier estimate of the median time from randomization to disease progression or death due to disease progression within the oxaliplatin stratum
Time Frame: Overall Study
Population: Intention-to-Treat
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | Oxaliplatin and Bevacizumab Plus Panitumumab | Oxaliplatin and Bevacizumab Without Panitumumab
Number analyzed (Participants) | 413 | 410
Month | 10.8 [9.5 to 11.3] | 11.4 [10.9 to 12.2]

5. Secondary Outcome: Time to Treatment Failure (Oxaliplatin)
Description: Kaplan-Meier estimate of the median time from randomization to the date the decision was made to discontinue treatment for a reason other than a complete response to treatment within the oxaliplatin stratum.
Time Frame: Overall study
Population: Intention-to-Treat
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | Oxaliplatin and Bevacizumab Plus Panitumumab | Oxaliplatin and Bevacizumab Without Panitumumab
Number analyzed (Participants) | 413 | 410
Month | 5.7 [5.5 to 6.0] | 5.9 [5.7 to 6.2]

6. Primary Outcome: Objective Tumor Response Through Week 12 (Irinotecan)
Description: Objective tumor response (complete or partial) rate through week 12 based on central review in the Irinotecan stratum
Time Frame: Overall Study
Population: Intention-to-Treat
Measure: Number; unit: Participant
Arm/Group | Irinotecan and Bevacizumab Plus Panitumumab | Irinotecan and Bevacizumab Without Panitumumab
Number analyzed (Participants) | 115 | 115
Participant | 29 | 27
Statistical Analysis 1: Comparison: Irinotecan and Bevacizumab Plus Panitumumab vs Irinotecan and Bevacizumab Without Panitumumab; Test type: Superiority or Other; p = 0.738, Regression, Logistic; Model covariates were ECOG status, prior adjuvant chemotherapy, number of metastatic organs, and primary disease site; Odds Ratio (OR) = 1.11, 95% CI [0.60 to 2.05]

7. Secondary Outcome: Overall Survival (Irinotecan)
Description: Incidence of mortality from any cause in groups treated with Irinotecan. Incidence is provided in lieu of the median time to death since the median or its measure of dispersion was not estimable for at least one treatment arm.
Time Frame: Overall study
Population: Intention-to-Treat
Measure: Number; unit: Participant
Arm/Group | Irinotecan and Bevacizumab Plus Panitumumab | Irinotecan and Bevacizumab Without Panitumumab
Number analyzed (Participants) | 115 | 115
Participant | 26 | 18
Statistical Analysis 1: Comparison: Irinotecan and Bevacizumab Plus Panitumumab vs Irinotecan and Bevacizumab Without Panitumumab; Test type: Superiority or Other; p = 0.257, Regression, Cox; Model covariates were ECOG status, prior adjuvant chemotherapy, number of metastatic organs, and primary disease site; Hazard Ratio (HR) = 1.42, 95% CI [0.77 to 2.62]

8. Secondary Outcome: Progression-free Survival (Irinotecan)
Description: as for outcome 1
Time Frame: Overall Study
Population: Intention-to-Treat
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | Irinotecan and Bevacizumab Plus Panitumumab | Irinotecan and Bevacizumab Without Panitumumab
Number analyzed (Participants) | 115 | 115
Month | 10.1 [8.2 to 13.7] | 11.7 [9.0 to 13.2]

9. Post Hoc Outcome: Progression-free Survival (Wild-type KRAS)
Description: Kaplan-Meier estimate of the median time from randomization to death from any cause or first observed disease progression in groups treated with oxaliplatin and having a wild-type Kirsten Rat Sarcoma Virus Oncogene (KRAS)
Time Frame: Overall Study
Population: Subset of the KRAS Efficacy Analysis Set, composed of participants from the intention-to-treat set who received at least 1 dose of first-line treatment and for whom KRAS mutation status was assessed as wild-type, who were treated with oxaliplatin
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | Oxaliplatin and Bevacizumab Plus Panitumumab | Oxaliplatin and Bevacizumab Without Panitumumab
Number analyzed (Participants) | 201 | 203
Month | 9.8 [8.4 to 11.3] | 11.5 [10.6 to 12.3]
Statistical Analysis 1: Comparison: Oxaliplatin and Bevacizumab Plus Panitumumab vs Oxaliplatin and Bevacizumab Without Panitumumab; Test type: Superiority or Other; Hazard Ratio (HR) = 1.36, 95% CI [1.04 to 1.77]

10. Post Hoc Outcome: Progression-free Survival (Mutant KRAS)
Description: Kaplan-Meier estimate of the median time from randomization to death from any cause or first observed disease progression in groups treated with oxaliplatin and having a mutant Kirsten Rat Sarcoma Virus Oncogene (KRAS)
Time Frame: Overall Study
Population: Subset of the KRAS Efficacy Analysis Set, composed of participants from the intention-to-treat set who received at least 1 dose of first-line treatment and for whom KRAS mutation status was assessed as mutant, who were treated with oxaliplatin
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | Oxaliplatin and Bevacizumab Plus Panitumumab | Oxaliplatin and Bevacizumab Without Panitumumab
Number analyzed (Participants) | 135 | 125
Month | 10.4 [9.1 to 11.3] | 11.0 [9.9 to 12.8]
Statistical Analysis 1: Comparison: Oxaliplatin and Bevacizumab Plus Panitumumab vs Oxaliplatin and Bevacizumab Without Panitumumab; Test type: Superiority or Other; Hazard Ratio (HR) = 1.25, 95% CI [0.91 to 1.71]

11. Post Hoc Outcome: Overall Survival (Wild-type KRAS)
Description: Kaplan-Meier estimate of the median time from randomization to death from any cause in groups treated with Oxaliplatin and having a wild-type Kirsten Rat Sarcoma Virus Oncogene (KRAS). Since the measure of dispersion could not be estimated for at least one treatment arm, participant incidence is provided in lieu of the median
Time Frame: Overall Study
Population: as for outcome 9
Measure: Number; unit: Participant
Arm/Group | Oxaliplatin and Bevacizumab Plus Panitumumab | Oxaliplatin and Bevacizumab Without Panitumumab
Number analyzed (Participants) | 201 | 203
Participant | 71 | 46
Statistical Analysis 1: Comparison: Oxaliplatin and Bevacizumab Plus Panitumumab vs Oxaliplatin and Bevacizumab Without Panitumumab; Test type: Superiority or Other; Hazard Ratio (HR) = 1.89, 95% CI [1.30 to 2.75]

12. Post Hoc Outcome: Overall Survival (Mutant KRAS)
Description: Kaplan-Meier estimate of the median time from randomization to death from any cause in groups treated with Oxaliplatin and having a mutant Kirsten Rat Sarcoma Virus Oncogene (KRAS). Since the measure of dispersion could not be estimated for at least one treatment arm, participant incidence is provided in lieu of the median.
Time Frame: Overall Study
Population: as for outcome 10
Measure: Number; unit: Participant
Arm/Group | Oxaliplatin and Bevacizumab Plus Panitumumab | Oxaliplatin and Bevacizumab Without Panitumumab
Number analyzed (Participants) | 135 | 125
Participant | 47 | 45
Statistical Analysis 1: Comparison: Oxaliplatin and Bevacizumab Plus Panitumumab vs Oxaliplatin and Bevacizumab Without Panitumumab; Test type: Superiority or Other; Hazard Ratio (HR) = 1.02, 95% CI [0.67 to 1.54]

13. Post Hoc Outcome: Objective Tumor Response Rate (Wild-type KRAS)
Description: Best overall response of complete or partial response in participants treated with irinotecan and having a wild-type Kirsten Rat Sarcoma Virus Oncogene (KRAS)
Time Frame: Overall Study
Population: Subset of the KRAS Efficacy Analysis Set, composed of participants from the intention-to-treat set who received at least 1 dose of first-line treatment and for whom KRAS mutation status was assessed as wild-type, who were treated with irinotecan
Measure: Number; unit: Participant
Arm/Group | Irinotecan and Bevacizumab Plus Panitumumab | Irinotecan and Bevacizumab Without Panitumumab
Number analyzed (Participants) | 57 | 58
Participant | 31 | 28
Statistical Analysis 1: Comparison: Irinotecan and Bevacizumab Plus Panitumumab vs Irinotecan and Bevacizumab Without Panitumumab; Test type: Superiority or Other; Odds Ratio (OR) = 1.28, 95% CI [0.61 to 2.66]

14. Post Hoc Outcome: Objective Tumor Response Rate (Mutant KRAS)
Description: Best overall response of complete or partial response in participants treated with irinotecan and having a mutant Kirsten Rat Sarcoma Virus Oncogene (KRAS)
Time Frame: Overall Study
Population: Subset of the KRAS Efficacy Analysis Set, composed of participants from the intention-to-treat set who received at least 1 dose of first-line treatment and for whom KRAS mutation status was assessed as mutant, who were treated with irinotecan
Measure: Number; unit: Participant
Arm/Group | Irinotecan and Bevacizumab Plus Panitumumab | Irinotecan and Bevacizumab Without Panitumumab
Number analyzed (Participants) | 47 | 39
Participant | 14 | 15
Statistical Analysis 1: Comparison: Irinotecan and Bevacizumab Plus Panitumumab vs Irinotecan and Bevacizumab Without Panitumumab; Test type: Superiority or Other; Odds Ratio (OR) = 0.68, 95% CI [0.28 to 1.67]

15. Secondary Outcome: Objective Tumor Response Rate (Irinotecan)
Description: Best overall response of complete or partial response within irinotecan stratum
Time Frame: Overall Study
Population: Intention-to-Treat
Measure: Number; unit: Participant
Arm/Group | Irinotecan and Bevacizumab Plus Panitumumab | Irinotecan and Bevacizumab Without Panitumumab
Number analyzed (Participants) | 115 | 115
Participant | 49 | 46

16. Secondary Outcome: Time to Progression (Irinotecan)
Description: Kaplan-Meier estimate of the median time from randomization to disease progression or death due to disease progression within the irinotecan stratum
Time Frame: Overall Study
Population: Intention-to-Treat
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | Irinotecan and Bevacizumab Plus Panitumumab | Irinotecan and Bevacizumab Without Panitumumab
Number analyzed (Participants) | 115 | 115
Month | 11.1 [8.3 to 14.1] | 11.9 [9.0 to 13.2]

17. Secondary Outcome: Time to Treatment Failure (Irinotecan)
Description: Kaplan-Meier estimate of the median time from randomization to the date the decision was made to discontinue treatment for a reason other than a complete response to treatment within the irinotecan stratum
Time Frame: Overall Study
Population: Intention-to-Treat
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | Irinotecan and Bevacizumab Plus Panitumumab | Irinotecan and Bevacizumab Without Panitumumab
Number analyzed (Participants) | 115 | 115
Month | 6.6 [5.9 to 8.0] | 6.0 [4.8 to 6.9]

ADVERSE EVENTS:
Time Frame: First dose through maximum of safety FU or 30 days after last dose
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Panit. Plus Bevacizumab With Chemotherapy | Bevacizumab With Chemotherapy
Serious Adverse Events (participants affected / at risk) | 306/518 | 188/510
Other Adverse Events (participants affected / at risk) | 516/518 | 505/510
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panit. Plus Bevacizumab With Chemotherapy (N=518) | Bevacizumab With Chemotherapy (N=510)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 4
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 20 | 9
GRANULOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 1
HAEMOLYSIS (Blood and lymphatic system disorders) | 0 | 1
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 | 1
LEUKOPENIA (Blood and lymphatic system disorders) | 3 | 2
NEUTROPENIA (Blood and lymphatic system disorders) | 9 | 8
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 | 1
SPLENIC INFARCTION (Blood and lymphatic system disorders) | 1 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 6 | 5
ANGINA PECTORIS (Cardiac disorders) | 3 | 5
ANGINA UNSTABLE (Cardiac disorders) | 1 | 0
ARRHYTHMIA (Cardiac disorders) | 2 | 2
ARTERIOSPASM CORONARY (Cardiac disorders) | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 3 | 2
ATRIAL FLUTTER (Cardiac disorders) | 0 | 1
CARDIAC ARREST (Cardiac disorders) | 3 | 1
CARDIAC FAILURE (Cardiac disorders) | 0 | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 3 | 4
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 2 | 1
CARDIOMYOPATHY (Cardiac disorders) | 1 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 | 2
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 4
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 1 | 0
PALPITATIONS (Cardiac disorders) | 1 | 1
PERICARDIAL EFFUSION (Cardiac disorders) | 2 | 0
SINUS TACHYCARDIA (Cardiac disorders) | 2 | 0
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 2 | 1
TACHYCARDIA (Cardiac disorders) | 2 | 1
VENTRICULAR FIBRILLATION (Cardiac disorders) | 1 | 0
DIPLOPIA (Eye disorders) | 1 | 0
ECTROPION (Eye disorders) | 1 | 0
EYELID DISORDER (Eye disorders) | 1 | 0
EYELID FUNCTION DISORDER (Eye disorders) | 1 | 0
VISUAL DISTURBANCE (Eye disorders) | 0 | 1
ABDOMINAL ADHESIONS (Gastrointestinal disorders) | 1 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 23 | 17
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 3 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 1
ANAL FISTULA (Gastrointestinal disorders) | 0 | 2
ANO-RECTAL ULCER (Gastrointestinal disorders) | 0 | 1
ASCITES (Gastrointestinal disorders) | 1 | 0
CAECITIS (Gastrointestinal disorders) | 1 | 0
COLITIS (Gastrointestinal disorders) | 4 | 2
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 1 | 1
COLITIS ULCERATIVE (Gastrointestinal disorders) | 1 | 0
COLONIC OBSTRUCTION (Gastrointestinal disorders) | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 4 | 1
CROHN'S DISEASE (Gastrointestinal disorders) | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 63 | 15
DIARRHOEA HAEMORRHAGIC (Gastrointestinal disorders) | 1 | 0
DIVERTICULAR PERFORATION (Gastrointestinal disorders) | 1 | 0
DUODENAL PERFORATION (Gastrointestinal disorders) | 1 | 0
DUODENAL ULCER PERFORATION (Gastrointestinal disorders) | 0 | 1
DUODENITIS (Gastrointestinal disorders) | 1 | 0
DYSPEPSIA (Gastrointestinal disorders) | 0 | 2
DYSPHAGIA (Gastrointestinal disorders) | 1 | 1
ENTERITIS (Gastrointestinal disorders) | 5 | 0
ENTEROCOLITIS (Gastrointestinal disorders) | 2 | 0
ENTEROCUTANEOUS FISTULA (Gastrointestinal disorders) | 1 | 0
ENTEROVESICAL FISTULA (Gastrointestinal disorders) | 0 | 1
EROSIVE OESOPHAGITIS (Gastrointestinal disorders) | 1 | 0
FAECALOMA (Gastrointestinal disorders) | 1 | 0
GASTRIC ULCER (Gastrointestinal disorders) | 1 | 1
GASTRIC ULCER PERFORATION (Gastrointestinal disorders) | 0 | 1
GASTROINTESTINAL FISTULA (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 7 | 4
GASTROINTESTINAL INFLAMMATION (Gastrointestinal disorders) | 0 | 1
GASTROINTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 2 | 0
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL PERFORATION (Gastrointestinal disorders) | 2 | 0
GASTROINTESTINAL TOXICITY (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL ULCER (Gastrointestinal disorders) | 1 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 3 | 0
HAEMATEMESIS (Gastrointestinal disorders) | 1 | 0
HAEMATOCHEZIA (Gastrointestinal disorders) | 1 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 1 | 0
ILEUS (Gastrointestinal disorders) | 7 | 3
ILEUS PARALYTIC (Gastrointestinal disorders) | 1 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 7 | 5
INTESTINAL PERFORATION (Gastrointestinal disorders) | 4 | 0
LARGE INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 3 | 1
MALLORY-WEISS SYNDROME (Gastrointestinal disorders) | 0 | 1
NAUSEA (Gastrointestinal disorders) | 24 | 7
OESOPHAGITIS (Gastrointestinal disorders) | 1 | 0
PANCREATITIS (Gastrointestinal disorders) | 1 | 1
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1 | 1
PERITONITIS (Gastrointestinal disorders) | 2 | 0
PNEUMOPERITONEUM (Gastrointestinal disorders) | 1 | 0
PROCTALGIA (Gastrointestinal disorders) | 0 | 2
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 2 | 2
RETROPERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 12 | 8
STOMATITIS (Gastrointestinal disorders) | 1 | 0
VOMITING (Gastrointestinal disorders) | 27 | 10
ASTHENIA (General disorders) | 10 | 4
CATHETER RELATED COMPLICATION (General disorders) | 2 | 1
CHEST PAIN (General disorders) | 1 | 1
CHILLS (General disorders) | 2 | 1
DISEASE PROGRESSION (General disorders) | 0 | 1
FATIGUE (General disorders) | 2 | 2
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 | 1
INFUSION RELATED REACTION (General disorders) | 0 | 1
MUCOSAL INFLAMMATION (General disorders) | 6 | 1
MULTI-ORGAN FAILURE (General disorders) | 1 | 0
NON-CARDIAC CHEST PAIN (General disorders) | 4 | 2
OEDEMA PERIPHERAL (General disorders) | 1 | 0
PAIN (General disorders) | 4 | 0
PELVIC MASS (General disorders) | 1 | 0
PNEUMATOSIS (General disorders) | 1 | 0
PYREXIA (General disorders) | 16 | 9
SWELLING (General disorders) | 1 | 0
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 2 | 0
ULCER (General disorders) | 1 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 1
GALLBLADDER FISTULA (Hepatobiliary disorders) | 1 | 0
HEPATIC FAILURE (Hepatobiliary disorders) | 1 | 0
HEPATIC LESION (Hepatobiliary disorders) | 0 | 1
JAUNDICE CHOLESTATIC (Hepatobiliary disorders) | 0 | 1
LIVER DISORDER (Hepatobiliary disorders) | 0 | 1
ANAPHYLACTIC REACTION (Immune system disorders) | 1 | 2
DRUG HYPERSENSITIVITY (Immune system disorders) | 2 | 1
HYPERSENSITIVITY (Immune system disorders) | 4 | 1
ABDOMINAL ABSCESS (Infections and infestations) | 2 | 0
ABDOMINAL INFECTION (Infections and infestations) | 1 | 0
ABSCESS (Infections and infestations) | 2 | 0
ACUTE SINUSITIS (Infections and infestations) | 1 | 0
APPENDICITIS (Infections and infestations) | 0 | 1
BACTERAEMIA (Infections and infestations) | 5 | 4
BACTERIAL INFECTION (Infections and infestations) | 1 | 0
BACTERIAL SEPSIS (Infections and infestations) | 2 | 0
BRONCHITIS (Infections and infestations) | 0 | 3
CANDIDIASIS (Infections and infestations) | 1 | 1
CATHETER RELATED INFECTION (Infections and infestations) | 7 | 2
CATHETER SEPSIS (Infections and infestations) | 0 | 1
CELLULITIS (Infections and infestations) | 4 | 1
CELLULITIS GANGRENOUS (Infections and infestations) | 1 | 0
CELLULITIS STAPHYLOCOCCAL (Infections and infestations) | 2 | 0
CLOSTRIDIAL INFECTION (Infections and infestations) | 3 | 1
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 1 | 0
CYSTITIS KLEBSIELLA (Infections and infestations) | 0 | 1
DEVICE RELATED INFECTION (Infections and infestations) | 1 | 1
DIVERTICULITIS (Infections and infestations) | 0 | 1
ESCHERICHIA BACTERAEMIA (Infections and infestations) | 1 | 0
EXTRADURAL ABSCESS (Infections and infestations) | 1 | 0
FUNGAEMIA (Infections and infestations) | 0 | 1
FUNGAL INFECTION (Infections and infestations) | 1 | 0
FUNGAL SEPSIS (Infections and infestations) | 1 | 0
FUNGAL SKIN INFECTION (Infections and infestations) | 1 | 1
GASTROENTERITIS (Infections and infestations) | 4 | 3
GASTROENTERITIS VIRAL (Infections and infestations) | 1 | 0
HERPES SIMPLEX (Infections and infestations) | 1 | 0
INFECTION (Infections and infestations) | 2 | 1
INTERTRIGO CANDIDA (Infections and infestations) | 1 | 0
INTERVERTEBRAL DISCITIS (Infections and infestations) | 1 | 0
KIDNEY INFECTION (Infections and infestations) | 1 | 0
MEDIASTINITIS (Infections and infestations) | 1 | 0
MENINGITIS CRYPTOCOCCAL (Infections and infestations) | 0 | 1
MUSCLE ABSCESS (Infections and infestations) | 0 | 1
NECROTISING FASCIITIS (Infections and infestations) | 2 | 0
NEUTROPENIC INFECTION (Infections and infestations) | 1 | 0
NEUTROPENIC SEPSIS (Infections and infestations) | 1 | 0
OSTEOMYELITIS (Infections and infestations) | 1 | 1
PAROTITIS (Infections and infestations) | 1 | 0
PELVIC ABSCESS (Infections and infestations) | 2 | 0
PERIRECTAL ABSCESS (Infections and infestations) | 2 | 0
PERITONEAL INFECTION (Infections and infestations) | 1 | 0
PERITONITIS BACTERIAL (Infections and infestations) | 1 | 0
PNEUMONIA (Infections and infestations) | 3 | 9
PNEUMONIA BACTERIAL (Infections and infestations) | 1 | 0
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 1 | 1
PYELONEPHRITIS (Infections and infestations) | 2 | 1
RASH PUSTULAR (Infections and infestations) | 1 | 0
RECTAL ABSCESS (Infections and infestations) | 0 | 1
RETROPERITONEAL ABSCESS (Infections and infestations) | 2 | 0
SEPSIS (Infections and infestations) | 16 | 8
SEPTIC SHOCK (Infections and infestations) | 2 | 3
SINUSITIS (Infections and infestations) | 0 | 1
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 3 | 1
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 | 1
STREPTOCOCCAL BACTERAEMIA (Infections and infestations) | 0 | 1
TRACHEOBRONCHITIS (Infections and infestations) | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 7 | 2
URINARY TRACT INFECTION FUNGAL (Infections and infestations) | 1 | 0
UROSEPSIS (Infections and infestations) | 2 | 1
WOUND INFECTION (Infections and infestations) | 3 | 0
ANASTOMOTIC LEAK (Injury, poisoning and procedural complications) | 1 | 0
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 0 | 1
CARBON MONOXIDE POISONING (Injury, poisoning and procedural complications) | 0 | 1
CONTUSION (Injury, poisoning and procedural complications) | 2 | 0
DRUG TOXICITY (Injury, poisoning and procedural complications) | 0 | 1
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 1
FOOT FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
GASTROINTESTINAL STOMA COMPLICATION (Injury, poisoning and procedural complications) | 0 | 1
HIP FRACTURE (Injury, poisoning and procedural complications) | 3 | 0
IMPLANTABLE DEFIBRILLATOR MALFUNCTION (Injury, poisoning and procedural complications) | 1 | 0
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 | 1
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1 | 0
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 2
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
WOUND (Injury, poisoning and procedural complications) | 1 | 0
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 1 | 1
BLOOD AMYLASE INCREASED (Investigations) | 0 | 1
BLOOD MAGNESIUM DECREASED (Investigations) | 0 | 1
BLOOD POTASSIUM DECREASED (Investigations) | 1 | 0
ELECTROCARDIOGRAM ABNORMAL (Investigations) | 1 | 0
HAEMOGLOBIN INCREASED (Investigations) | 1 | 0
LIPASE INCREASED (Investigations) | 0 | 1
NEUTROPHIL COUNT DECREASED (Investigations) | 1 | 1
PLATELET COUNT DECREASED (Investigations) | 1 | 1
PROTHROMBIN TIME PROLONGED (Investigations) | 1 | 0
WEIGHT DECREASED (Investigations) | 2 | 0
ACIDOSIS (Metabolism and nutrition disorders) | 1 | 0
ANOREXIA (Metabolism and nutrition disorders) | 5 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 72 | 21
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 0 | 1
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 2 | 1
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 0 | 1
GOUT (Metabolism and nutrition disorders) | 0 | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 2 | 0
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 2 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 12 | 4
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 6 | 0
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 3 | 1
MALNUTRITION (Metabolism and nutrition disorders) | 0 | 1
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 1 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5 | 6
FISTULA (Musculoskeletal and connective tissue disorders) | 2 | 0
INTERVERTEBRAL DISC DEGENERATION (Musculoskeletal and connective tissue disorders) | 0 | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 3 | 0
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 | 2
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 1
SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 2 | 0
SOFT TISSUE NECROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 | 4
COLON CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 2
COLORECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
COLORECTAL CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
HEPATIC NEOPLASM MALIGNANT RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
APHASIA (Nervous system disorders) | 0 | 1
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 | 1
CEREBRAL ISCHAEMIA (Nervous system disorders) | 1 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 0
CONVULSION (Nervous system disorders) | 5 | 1
COORDINATION ABNORMAL (Nervous system disorders) | 1 | 0
DIZZINESS (Nervous system disorders) | 3 | 4
ENCEPHALOPATHY (Nervous system disorders) | 0 | 1
GRAND MAL CONVULSION (Nervous system disorders) | 1 | 0
HEADACHE (Nervous system disorders) | 3 | 3
HYPERTENSIVE ENCEPHALOPATHY (Nervous system disorders) | 0 | 1
LETHARGY (Nervous system disorders) | 1 | 0
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 | 1
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 1 | 0
NEUROPATHY (Nervous system disorders) | 1 | 0
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 | 1
RADICULOPATHY (Nervous system disorders) | 0 | 1
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 0 | 1
SYNCOPE (Nervous system disorders) | 3 | 3
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 3 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 2 | 0
DEPRESSION (Psychiatric disorders) | 2 | 0
MAJOR DEPRESSION (Psychiatric disorders) | 1 | 0
MENTAL STATUS CHANGES (Psychiatric disorders) | 1 | 1
PANIC ATTACK (Psychiatric disorders) | 1 | 0
SUICIDE ATTEMPT (Psychiatric disorders) | 1 | 0
CALCULUS URINARY (Renal and urinary disorders) | 0 | 1
DYSURIA (Renal and urinary disorders) | 1 | 0
FAECALURIA (Renal and urinary disorders) | 0 | 1
HAEMATURIA (Renal and urinary disorders) | 1 | 1
HYDRONEPHROSIS (Renal and urinary disorders) | 2 | 0
NEPHROLITHIASIS (Renal and urinary disorders) | 2 | 0
RENAL FAILURE (Renal and urinary disorders) | 6 | 2
RENAL FAILURE ACUTE (Renal and urinary disorders) | 2 | 4
URETERIC OBSTRUCTION (Renal and urinary disorders) | 1 | 0
URETHRAL OBSTRUCTION (Renal and urinary disorders) | 1 | 0
URINARY RETENTION (Renal and urinary disorders) | 1 | 0
URINARY TRACT PAIN (Renal and urinary disorders) | 1 | 0
VESICAL FISTULA (Renal and urinary disorders) | 1 | 0
FEMALE GENITAL TRACT FISTULA (Reproductive system and breast disorders) | 1 | 2
VULVAL DISORDER (Reproductive system and breast disorders) | 1 | 0
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 3 | 0
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 2
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 1 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 1
DYSAESTHESIA PHARYNX (Respiratory, thoracic and mediastinal disorders) | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 8 | 12
DYSPNOEA EXACERBATED (Respiratory, thoracic and mediastinal disorders) | 1 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 2 | 0
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 3 | 1
PLATYPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 3 | 1
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 2 | 0
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 2
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 35 | 17
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 1
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 2 | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 1
DERMATITIS (Skin and subcutaneous tissue disorders) | 1 | 0
INTERTRIGO (Skin and subcutaneous tissue disorders) | 1 | 0
PETECHIAE (Skin and subcutaneous tissue disorders) | 0 | 1
PURPURA (Skin and subcutaneous tissue disorders) | 0 | 1
RASH (Skin and subcutaneous tissue disorders) | 5 | 0
SKIN REACTION (Skin and subcutaneous tissue disorders) | 1 | 0
TELANGIECTASIA (Skin and subcutaneous tissue disorders) | 1 | 0
COLECTOMY (Surgical and medical procedures) | 2 | 0
CRYOTHERAPY (Surgical and medical procedures) | 0 | 1
HEPATECTOMY (Surgical and medical procedures) | 14 | 6
HEPATIC EMBOLISATION (Surgical and medical procedures) | 0 | 1
HIGH FREQUENCY ABLATION (Surgical and medical procedures) | 2 | 1
LESION EXCISION (Surgical and medical procedures) | 1 | 0
LIVER OPERATION (Surgical and medical procedures) | 0 | 1
LUNG NEOPLASM SURGERY (Surgical and medical procedures) | 0 | 1
ARTERIOSCLEROSIS (Vascular disorders) | 1 | 0
AXILLARY VEIN THROMBOSIS (Vascular disorders) | 1 | 1
CIRCULATORY COLLAPSE (Vascular disorders) | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 17 | 12
EMBOLISM (Vascular disorders) | 1 | 1
HAEMATOMA (Vascular disorders) | 2 | 2
HAEMORRHAGE (Vascular disorders) | 0 | 1
HYPERTENSION (Vascular disorders) | 4 | 5
HYPOTENSION (Vascular disorders) | 4 | 6
JUGULAR VEIN THROMBOSIS (Vascular disorders) | 1 | 1
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 1 | 0
SUBCLAVIAN VEIN THROMBOSIS (Vascular disorders) | 2 | 2
THROMBOSIS (Vascular disorders) | 3 | 2
VENA CAVA THROMBOSIS (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Panit. Plus Bevacizumab With Chemotherapy (N=518) | Bevacizumab With Chemotherapy (N=510)
ANAEMIA (Blood and lymphatic system disorders) | 177 | 147
LEUKOPENIA (Blood and lymphatic system disorders) | 53 | 60
NEUTROPENIA (Blood and lymphatic system disorders) | 179 | 207
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 71 | 108
CONJUNCTIVITIS (Eye disorders) | 31 | 6
LACRIMATION INCREASED (Eye disorders) | 34 | 34
VISION BLURRED (Eye disorders) | 29 | 22
ABDOMINAL PAIN (Gastrointestinal disorders) | 132 | 114
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 48 | 38
CONSTIPATION (Gastrointestinal disorders) | 217 | 187
DIARRHOEA (Gastrointestinal disorders) | 385 | 350
DRY MOUTH (Gastrointestinal disorders) | 30 | 31
DYSPEPSIA (Gastrointestinal disorders) | 86 | 72
DYSPHAGIA (Gastrointestinal disorders) | 31 | 18
FLATULENCE (Gastrointestinal disorders) | 33 | 48
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 35 | 40
HAEMORRHOIDS (Gastrointestinal disorders) | 41 | 49
NAUSEA (Gastrointestinal disorders) | 359 | 368
ORAL PAIN (Gastrointestinal disorders) | 46 | 40
PROCTALGIA (Gastrointestinal disorders) | 34 | 24
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 43 | 34
STOMATITIS (Gastrointestinal disorders) | 171 | 91
VOMITING (Gastrointestinal disorders) | 215 | 199
ASTHENIA (General disorders) | 92 | 68
CHILLS (General disorders) | 63 | 55
FATIGUE (General disorders) | 354 | 371
MUCOSAL INFLAMMATION (General disorders) | 159 | 104
OEDEMA PERIPHERAL (General disorders) | 54 | 61
PAIN (General disorders) | 38 | 39
PYREXIA (General disorders) | 111 | 82
TEMPERATURE INTOLERANCE (General disorders) | 65 | 99
PARONYCHIA (Infections and infestations) | 51 | 0
SINUSITIS (Infections and infestations) | 26 | 35
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 26 | 38
URINARY TRACT INFECTION (Infections and infestations) | 72 | 47
NEUTROPHIL COUNT DECREASED (Investigations) | 25 | 32
WEIGHT DECREASED (Investigations) | 166 | 107
ANOREXIA (Metabolism and nutrition disorders) | 211 | 155
DECREASED APPETITE (Metabolism and nutrition disorders) | 50 | 51
DEHYDRATION (Metabolism and nutrition disorders) | 129 | 72
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 43 | 34
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 35 | 9
HYPOKALAEMIA (Metabolism and nutrition disorders) | 172 | 73
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 148 | 14
HYPONATRAEMIA (Metabolism and nutrition disorders) | 26 | 12
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 60 | 71
BACK PAIN (Musculoskeletal and connective tissue disorders) | 71 | 74
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 30 | 31
MYALGIA (Musculoskeletal and connective tissue disorders) | 29 | 46
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 54 | 49
SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 33 | 40
DIZZINESS (Nervous system disorders) | 107 | 93
DYSGEUSIA (Nervous system disorders) | 95 | 97
HEADACHE (Nervous system disorders) | 95 | 113
HYPOAESTHESIA (Nervous system disorders) | 33 | 41
NEUROPATHY (Nervous system disorders) | 98 | 115
NEUROPATHY PERIPHERAL (Nervous system disorders) | 94 | 106
PARAESTHESIA (Nervous system disorders) | 82 | 104
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 64 | 85
ANXIETY (Psychiatric disorders) | 61 | 65
DEPRESSION (Psychiatric disorders) | 91 | 68
INSOMNIA (Psychiatric disorders) | 122 | 126
HAEMATURIA (Renal and urinary disorders) | 29 | 23
PROTEINURIA (Renal and urinary disorders) | 46 | 46
COUGH (Respiratory, thoracic and mediastinal disorders) | 106 | 97
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 31 | 31
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 126 | 100
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 146 | 164
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 27 | 38
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 71 | 57
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 26 | 25
ALOPECIA (Skin and subcutaneous tissue disorders) | 111 | 86
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 179 | 7
DRY SKIN (Skin and subcutaneous tissue disorders) | 143 | 38
ERYTHEMA (Skin and subcutaneous tissue disorders) | 75 | 24
EXFOLIATIVE RASH (Skin and subcutaneous tissue disorders) | 33 | 2
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 41 | 17
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 52 | 31
PRURITUS (Skin and subcutaneous tissue disorders) | 141 | 33
RASH (Skin and subcutaneous tissue disorders) | 331 | 71
SKIN FISSURES (Skin and subcutaneous tissue disorders) | 72 | 10
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 13 | 26
SKIN ULCER (Skin and subcutaneous tissue disorders) | 32 | 5
DEEP VEIN THROMBOSIS (Vascular disorders) | 26 | 25
HYPERTENSION (Vascular disorders) | 86 | 107
HYPOTENSION (Vascular disorders) | 49 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multi-center studies, the investigator agrees not to publish any results before the first multi-center publication.